CLINICAL TRIAL: NCT04959084
Title: Effectiveness of Laser Acupuncture and Pelvic Floor Training on Stress Urinary Incontinence in Obese Postmenopausal Women
Brief Title: Laser Acupuncture and Pelvic Floor Training on Stress Urinary Incontinence Postmenopausal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Mohamed Aly Embaby, Assistant professor for physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LA and PFT in SUI
Record Dates: First submitted 2021-06-28; First posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Stress; Urinary; Incontinence
Keywords: laser acupuncture; pelvic floor training; Urinary incontinence; postmenopausal
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Experimental): Acupuncture group A , consisting of 20 women will be received laser acupuncture therapy and pelvic floor training every other day for 30 min , 3 times per week for 12 sessions
  Interventions: Other: Laser acupuncture therapy and pelvic floor training
- Medical (No Intervention): Medical group B, consisting of 20 women will be maintained their ordinary medical treatment

INTERVENTIONS:
Other: Laser acupuncture therapy and pelvic floor training — The laser will be applied directly to the skin over acupuncture points and each point receive a shoot of 65 seconds followed by Pelvic floor exercises for 15 min.
  Arms: Acupuncture

SUMMARY:
This study will be directed to determine the effectiveness of laser acupuncture(LA) and pelvic floor training (PFT) on stress urinary incontinence (SUI) in obese postmenopausal women. Forty obese postmenopausal women will be selected , suffering from mild to moderate stress urinary incontinence from mild to moderate stress urinary incontinence, their age ranges from 50-65 years old and the body mass index (BMI) ≥ 30 ≤ 40 Kg/m2. then separate randomly into two equivalent gatherings. The study group (A) will receive laser acupuncture therapy and pelvic floor training for 30 min every other day for 12 sessions (3 times per week). While the control group (B) maintaining their ordinary medical treatment. All participants will be assessed the pelvic floor muscles strength by using Modified oxford grading scale and perineometer before starting intervention and at the end of the 12th session.

DETAILED DESCRIPTION:
Menopause is the most significant period in a woman's life and brings in many physiological changes that affect life permanently. There have been a lot of opinions about the symptoms that appear before, during and after the onset of menopause . Menopause is associated with weight gain, as well as an increase in hypertension and diabetes. Estrogen deficiency can cause hormonal changes that contribute to the development of osteoporosis. Menopause is marked by hot flushes, sweating (especially at night), irritability, concentration issues, joint pain, vaginal dryness, and urogenital disorders( high rate of incontinence) .

Postmenopausal women are at danger for urogynecology dysfunction, incontinence, prolapse, and sexual dysfunction as circulating estrogen levels decrease with age. Their signs and symptoms may have a big impact on one's personal satisfaction. Menopause occurs at a normal age of 51 years in women, with the majority of women experiencing it between the ages of 45 and 55. As a result, women should expect to live for another 30 years after menopause .

SUI affects 20-30% of young women, 30-40% of moderately aged women, and up to half of the women in their later years, making it a major social issue that influences the greater part of postmenopausal women. This issue significantly influences the personal satisfaction of influenced women , also urinary incontinence may affect the functional ability of elderly females. Stress urinary incontinence is the most widespread type of incontinence (SUI). According to a study, SUI is often associated with conditions that cause high intra-abdominal pressure, for example, pregnancy with or without vaginal conveyance, obesity, and difficult physical work. The urogenital tract and pelvic floor contain estrogen and progesterone receptors. This may mean that these hormones play a role in continence. Estrogen does, in fact, increase urethral closure pressure, possibly due to increased blood flow. Estrogen has also been shown to improve the epithelia in the vagina, urethra, and bladder wall in postmenopausal women. As a result, it is reasonable to assume that using postmenopausal hormone therapy (HT) would reduce the risk of SUI .

The most well-known and potentially modifiable danger factor for the advancement of UI is obesity. In some studies, a positive connection between UI and body mass index (BMI) has effectively been created. Weight has a direct dose effect on incontinence, with every 5-unit expansion in BMI raising the risk of incontinence by 20 to 70%. And compared to ordinary-weight patients, obese patients have about double the risk of presenting with UI. Increased intra-abdominal pressure, as well as constant tension on tendons and nerves, can bother or cause pelvic floor problems by causing excessive stretching [6]. Increased intra-abdominal pressure (IAP) caused by obesity stresses the pelvic floor and leads to the growth of SUI, according to the prevailing unifying theory.

Changes in one's lifestyle can help with simple stress incontinence. Weight loss, liquid restriction, expected voiding, Kegel muscle preparation, and biofeedback are among the modifications. In addition, there is a group of incontinence schemes that can be used .The aim of timed voiding is to keep the bladder from being too full. Exercises to strengthen the pelvic floor muscles can aid elderly women with urinary incontinence .

Although there are many ways to treat urinary incontinence such as drug treatment and surgical intervention, but physical therapy is one of the most successful and best treatment methods used with patients with urinary incontinence, this method it is the best treatment methods that help patients strengthen the pelvic muscles and get rid of urinary incontinence .

Incontinence is often treated with pelvic floor exercise (Kegel's Exercise). It consists of repeated contractions of the pelvic floor muscles, especially the pubococcygeus muscle, to strengthen the muscles and improve micturition control . Pelvic floor exercise, including how to do a Kegel press, can be shown to the patient. When contracting the muscles used to avoid the outflow of urine or flatus, keep the stomach and thighs relaxed . In addition to laser treatment has a major role in the treatment of many cases .

Low-intensity laser therapy (LILT) is a type of phototherapy utilized as a therapy for many conditions, including musculoskeletal and delicate tissue wounds and persistent ulceration. Such lasers additionally prescribed as a successful choice to metal needles for the incitement of acupuncture or musculoskeletal trigger focus. This type of treatment is ordinarily named "Laser Acupuncture" to recognize it from the more extensive restorative utilization of such laser gadgets .

Laser acupuncture is essentially safer than needle acupuncture because of the non- intrusive nature of treatment (for example in instances of disease) and a more suitable technique for the incitement of difficult points as auricular acupuncture points or points around the perineum or privates (e.g., for sexual dysfunction) . The lumbosacral area of the body may be treated with laser acupuncture to mimic pelvic floor muscles. Laser acupuncture can stimulate the posterior S1 via BL31, S2 via BL32, S3 via BL33, S4 via BL34, and the pudendal nerve via BL35 at the lumbosacral area, as these techniques are effective in treating SUI. As a result, laser acupuncture can aid in the reinnervation and strengthening of pelvic floor muscles, thereby alleviating SUI symptoms .

ELIGIBILITY:
Inclusion Criteria:

* Forty obese postmenopausal women suffer from mild to moderate stress urinary incontinence
* Their age ranges from 50-65 years old
* The body mass index (BMI) ≥ 30 ≤ 40 Kg/m2.

Exclusion Criteria:

* neuromuscular disorders
* Lumbar disc prolapse
* Gynaecological disorders
* Pacemakers
* Tumors
* Dermatological conditions
* Patient who take anticoagulant agents.

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal women with mild to moderate stress urinary incontinence will be included in the study
Enrollment: 45 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in the pelvic floor muscles strength | 4 weeks following the end of sessions
  Modified oxford grading scale (MOS) Via vaginal palpation, it was used to measure pelvic floor muscle strength. The strength of PFMS is graded on a scale of 0-5. subjective assessment

CONTACTS AND LOCATIONS:
Overall Officials: Heba Embaby, Ph.D., Principal Investigator — Cairo University CU
Locations (1):
- Faculty of physical therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No